Dear Sir/Madam,

First of all, thank you for your evaluation. After a second review, we concluded that the study design was observational.

In our study, the volunteers will not receive any intervention. They are only expected to complete the 6-meter walking speed and handgrip strength test.

In addition, their sociodemographic information will be asked.

The results obtained will be analyzed using the SPSS program.

Parametric methods will be used to measure values suitable for normal distribution. In accordance with parametric methods, the "Independent Sample-t" test (t-table value) will be used to compare the measurement values of two independent groups, and the "ANOVA" test (F-table value) will be used to compare the measurement values of three or more independent groups. The "Tukey" method will be applied for pairwise comparisons of variables with significant differences for three or more groups, considering the homogeneity of variances.

Non-parametric methods will be used for measurement values unsuitable for normal distribution. By non-parametric methods, the "Mann-Whitney U" test (Z-table value) will be used for comparing the measurement values of two independent groups, and the "Kruskal-Wallis H" test ( $\chi$ 2-table value) will be used for comparing the measurement values of three or more independent groups. Bonferroni correction was applied for pairwise comparisons of variables with significant differences for three or more groups.

In cases where two quantitative variables are suitable for normal distribution, the "Pearson" correlation coeficient will be. In cases where at least one variable is unsuitable for normal distribution, the "Spearman" correlation coeficient will be used.

If you have any additional requests or questions, we are happy to inform you that we will try to explain.

Yours sincerely